CLINICAL TRIAL: NCT03582761
Title: A Phase IV Clinical Trial for Efficacy Evaluation for Inactivated Vaccine (Vero Cell) Against EV71: A Multicenter， Case-control Study.
Brief Title: Efficacy Evaluation for Inactivated Vaccine (Vero Cell) Against EV71
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Wuhan Institute of Biological Products Co., Ltd (Industry); Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT048
Record Dates: First submitted 2018-06-08; First posted 2018-07-11 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2019-05

CONDITIONS: Hand, Foot and Mouth Disease
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 320U /0.5ml in children (Experimental): EV71 vaccine of 320U /0.5ml will be given to 40000 children aged 6-35 months old on day0,28
  Interventions: Biological: EV71 vaccine

INTERVENTIONS:
Biological: EV71 vaccine — EV71 vaccine of 320U /0.5ml will be given to 40000 children aged 6-35 months old on day0,28

SUMMARY:
This study is a multicenter, case-control phase IV clinical trial to evaluate the effectiveness of the EV71 vaccine. About 40000 children in the town aged 6-35 months will be recruited and vaccinated with EV71 vaccines, which account for 20-40% of the children aged 6-35 months in the areas. The subjects will be vaccinated with EV71 vaccine at day 0 and day 28. Other children of appropriate age in the town will choose voluntarily whether or not to be vaccinated with EV71 vaccine. All children's vaccination of EV71 vaccines will be recorded in the study areas and the coverage rate of EV71 vaccine in the town will be calculated. The vaccination is expected to complete before the epidemic peak of HFMD.

Surveillance of HFMD cases caused by EV71 will be conducted in hospitals of the study areas for 10-12 months, which cover a whole HFMD epidemic period. Throat and anal swabs will be collected from children with a clinically diagnosed HFMD for typing of human enteroviruses tested by PCR. The HFMD cases with EV71 positive will be recruited as cases, while those with EV71 negative will be recruited as test-negative controls. Besides, for each EV71-associated HFMD cases, the investigators will select 4 community controls mateced with each case for age, sex and residence.

ELIGIBILITY:
Inclusion Criteria:

For vaccination group：

* Healthy children aged 6-35 months
* Subjects who have been clinically judged to be healthy by the researcher after being asked about the medical history and related physical examination
* The subjects' guardians agree the requirements of the protocol and the relevant follow up visits
* The subjects' guardians agree and sign the informed consent

For case group：

* Aged from 6 to 47 months
* Clinical diagnosis of HFMD
* At least one throat swab or anal swab detected EV71 positive by PCR
* The subjects' guardians agree and sign the informed consent

For hospital control group：

* Aged from 6 to 47 months
* Clinical diagnosis of HFMD
* Throat swabs or anal swabs are positive for enterovirus and negative for EV71
* The subjects' guardians agree and sign the informed consent

For community control group：

* Aged from 6 to 47 months
* No clinically diagnosed HFMDs, and no fever, HFMD suspected symptoms, such as hand, foot and mouth herpes
* The same gender as the matched case
* The age is similar to that of matched case (for cases ≥ 12 months of age, the age difference is within ±3 months, for case < 12 months of age, the age difference is within ±30 days)
* Near the residence of the case (the same village or adjacent village)
* The subjects' guardians agree and sign the informed consent

Exclusion Criteria:

For vaccination group：

* Subject who has a medical history of HFMD caused by EV71 or has been vaccinated with EV71 vaccine
* Subject who is known to be allegric to the componets of the vaccine
* Subject with fever or acute diseases or at acute stage of chronic diseases
* Subject with severe chronic diseases and allergies
* Subject with thrombocytopenia or hemorrhagic diseases
* Subject who is receiving immunosuppressive therapy or with immunodeficiency
* Subject with uncontrolled epilepsy and other progressive neurological illness, such as Guillain-Barre syndrome.

Exclusion Criteria for the second dose:

* Have severe allergic reaction after first dose
* Have severe adverse reactions related to first dose
* Any situation meet the exclusion criteria stated in the exclusion criteria for first dose
* Acute infection or illness
* Other factors that are not suitable for clinical trials according to the judgment of researchers For case group：
* Unknown of EV71 vaccination history
* EV71 related disease occurred within 28 days after the first vaccination
* The place of residence is not included in the study areas

For hospital control group：

* Unknown of EV71 vaccination history
* A history of HFMD caused by EV71 or unknown HFMD related pathogen
* The place of residence is not included in the study areas
* For community control group：
* For community control group：

For community control group：

* Unknown of EV71 vaccination history
* A history of HFMD caused by EV71 or unknown HFMD related pathogen

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40000 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Odds ratio (OR) of the immunization of EV-A71 vaccine in cases vs control groups | within 12 months after completion of vaccination
  Cases are defined as eligible patients who tested positive for enteroviruse 71. For each case, we will select two groups of control children, including hospital test-negative control and community control. Logistic regression is performed to calculate the odds ratio (OR) of vaccination in cases vs each of the control groups.

SECONDARY OUTCOMES:
Incidence and severity of adverse reactions/adverse events in children aged 6-35 months after EV71 vaccine receiving. | 1 month after completion of vaccination
  Incidence and severity of adverse reactions/adverse events in children aged 6-35 months within 1 month after completion of vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Feng-Cai, Master, Principal Investigator — Jiangsu Provincial Center for Diseases Control and Prevention
Locations (2):
- China (2):
  - Hubei Provincial Center for Diseases Control and Prevention, Wuhan, Hubei
  - Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes will be made available within 6 months of study completion.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the sponsor. Requestors will be required to sign a Date Access Agreement.